CLINICAL TRIAL: NCT05171400
Title: A New Drug Delivery System - Silk Fibroin Film Loaded or Not With Insulin on Palatal Mucosa Wound Healing: in Vitro Study and a Randomized Clinical Trial.
Brief Title: A New Drug Delivery System - Silk Fibroin Film Loaded or Not With Insulin on Palatal Mucosa Wound Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEPJMF11
Record Dates: First submitted 2021-09-28; First posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Wound Healing; Insulin; Palate; Wound
Keywords: Wound Healing; Drug Delivery System; Insulin; Fibroin
MeSH Terms: conditions — Insulin Resistance; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This is a double-blind, parallel, superiority, randomized clinical trial with 3 months of follow-up.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (CG) (Sham Comparator): The palatal wound area will not receive any treatment
  Interventions: Procedure: Palatal Wound
- Blank Film Group (BF) (Experimental): The palatal wound area will receive silk fibroin film as a dressing
  Interventions: Procedure: Palatal Wound; Device: Palatal Wound treated with Silk Fibroin Film
- Insulin-loaded film (IF) (Experimental): The palatal wound area will receive an insulin-loaded silk fibroin film as a drug delivery system
  Interventions: Procedure: Palatal Wound; Device: Palatal Wound treated with Insulin-loaded Silk Fibroin Film

INTERVENTIONS:
Procedure: Palatal Wound — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive 4.0 silk sutures.
Device: Palatal Wound treated with Silk Fibroin Film — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive a silk fibroin film and 4.0 silk sutures.
  Arms: Blank Film Group (BF)
Device: Palatal Wound treated with Insulin-loaded Silk Fibroin Film — With the goal to harvest the free gingival graft (FGG), an 8mm diameter scalpel will be used to ensure standardized wounds. Thereafter, a 2-mm thick FGG will be removed. The wound area will receive a silk fibroin film loaded with insulin and 4.0 silk sutures.
  Arms: Insulin-loaded film (IF)

SUMMARY:
The aim of the present study is to evaluate using clinical, patient-centered, immunological, microbiological, and histological parameters, the effect of silk fibroin films loaded or not with insulin in the repair of palatal mucosa open wounds.

DETAILED DESCRIPTION:
There are several types of periodontal and peri-implant soft tissue defects that require surgical treatment to reestablishment function and aesthetics. Therefore, surgical procedures for the reconstruction of the gingival and peri-implant tissues are routinely performed. However, these procedures do not always have predictable outcomes, and problems with the wound healing process can occur, which can impair the outcomes. To overcome this problem, new materials, drugs, and devices have been used to improve the results of surgical procedures. The present study is a controlled clinical trial that will include seventy-five patients with an indication of anterior maxillary tooth extraction for ridge preservation. The ridge preservation will be performed and a free gingival graft harvest from the palatal mucosa will be used to seal the socket entrance. Thereafter, the palatal wound will be randomly assigned into 3 groups: Control Group (C; n=25): open wound on palatal mucosa that will receive no treatment. Blank Film Group (BF; n=25): open wound on palatal mucosa that will receive silk fibroin film as dressing. Insulin-loaded film (IF; n=25): open wound on palatal mucosa that will receive an insulin-loaded silk fibroin film as a delivery system. Clinical, immunological, histological, and microbiome parameters will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 18 years, systemically healthy, with good oral hygiene, assessed by plaque index and gingival index less than 25% (Ainamo, Bay, 1975);
* Patients with no morphological or pathological conditions on the palatine donor area;
* Patients who present indication for extraction and ridge preservation;
* The tooth included in the study, as well as, the adjacent teeth do not present loss of periodontal insertion;
* Patients who agreed to and sign the formal consent to participate in the study after receiving an explanation of risks and benefits from an individual who was not a member of the present study (Resolution no. 118 - May, 2012, and Ethics and Code of Professional Conduct in Dentistry - 118/12).

Exclusion Criteria:

* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, and diabetes, among others) that will contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers patients;
* Pregnant or lactating patients;
* Patients who had had periodontal surgery on the study area;
* Patients who presents opportunistic oral lesions, mainly colonized the palate region;
* Use of dental prosthesis with palatal cover;
* Thin palatal mucosa (~2.0mm).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-08-02 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in the Remaining wound healing (RWA) | 90 days.
  Photographs will be taken from palatal wound with brightness, distance, and angle standardized. A scale will be placed in the palate as a reference to measure the area. These photographs will be exported to an image software (Image J - NIH, Bethesda, USA), and the wound area will be measured in square millimeters (Dias et al., 2015).

SECONDARY OUTCOMES:
Tissue Thickness (TT) | 90 days
  Tissue thickness of palatine masticatory mucosa will be assessed by a Cone Beam Computed Tomographic (CBCT). In order to standardize the volume measures, the FGG harvested stent, made of 1 mm thick rigid acrylic plates in vacuum plasticizer with radiopaque material, will be used by the patient at the time of the CBCT image acquisition.
Epithelialization (E) | 90 days
  Wound will be colored with Replack (Dentisply - York, Pensilvânia - USA) and quantity measured by Image J program. Then, with the total area of the wound, the epithelization % will be calculated (Ozcelik et al. 2008).
Early- wound healing index (EWHI) | 14 days
  According to Fickl et al. 2014 any modification in wound healing will be evaluated in five different degrees:
  * Complete wound closure with an absence of fibrin on the palate;
  * Complete wound closure with the presence of a fibrin line on palate;
  * Complete wound closure with the presence of a clot with fibrin on palate
  * Incomplete wound closure with partial tissue necrosis on palate;
  * Incomplete wound closure with total tissue necrosis on palate
Tissue Edema (TE) | 7 days
  Tissue edema will be evaluated with the score: 1 = absent; 2 = slight; 3 = moderate; or 4 = severe (Sanz-Moliner et, 2013).
Oral Health Impact Profile | 14 days
  Will be evaluated from a questionnaire with 14 questions based on 7 domains: functional limitations, physical pain, psychological discomfort, physical disability, psychological deficiency and social deficiency. The patient should respond to the questions within 14 days after the surgical procedure, performing a postoperative diary. For each question an answer must be given, represented in numbers, being: 0- Never; 1- Almost never; 2-Occasionally; 3-Quite frequent; 4-Very common; 5-I do not know (Tonetti MS et al. 2017)
Number of analgesics | 14 days
  Number of analgesics used during 14 days after the procedure will be reported at the same postoperative diary (Tonetti et al. 2017).
Patient Discomfort | 14 days
  By a visual analogic scale (VAS) of 100 mm to assess discomfort, patients will report pain diary during the 14 days after surgery. Scale extremes will be "no pain" to "extreme." (Tonetti et al. 2017).
Qualitative somatosensory testing (QualST) | 14 days
  This analysis will evaluate somatosensorial profiles and pain conditions. For this, different stimulus will be performed on the wound and the following tests will be applied: (1) Touch stimulus will be applied with a swab by a single application for 1-2 sec in the wound; (2) Cold stimulus will be applied by a stainless steel dental spatula (kept cool in ice water, approximately 0 °C) with wound direct contact during 1-2 sec; (3) The pinprick stimulus will be performed with a periodontal probe with moderate force on the wound area for 1-2 s (Baad-Hansen et al, 2013) Patient will report hypersensitivity, hyposensitivity, or normosensitivity to touch, cold and painful stimulus.
Immunologic Analysis | 7 days
  With the goal to obtain baseline data for this parameter, crevicular gingival fluid from the gingival area next to the donor area will be collected previous surgery. An absorbent paper (PerioPaper, Oraflow, Plainview, NY, EUA) will be placed at wound edges without pressure during 40s. Collects with blood contamination will be discarded. Samples will be stored into a sterilized Eppendorf containing 100 μL Phosphate Buffer Saline 0.05% Tween 2 (PBS) at - 80 C. Growth factors (VEGF and EGF), chemokines (MIP-1α, MCP-1α), and cytokines (IL1β, IL6, IL10, TNFα) levels will be determinate by the multiplex assay. Moreover, MMP-2, MMP-9, TIMP-1, TIMP-2 will be measured by the same commercial human commercial kit.
Histological Analysis | 180 days
  CTG will be harvested from the palatal area, the same area that received FGG protocol previously, using the same harvesting stent, during implant therapy. After CTG be harvested, a 2-mm thick will be removed from the graft (Azar et al., 2019) to perform biopsy analysis aiming to observe histological changes during healing process by previously use of silk fibroin film, charged or not with insulin, and spontaneous repair. The specimens will be immersed in 10% formalin for histological analysis which will be stained with hematoxylin-eosin and Masson's trichrome.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Study Director — Sao Paulo State University - Brazil; Manuela Maria V Miguel, MS, Principal Investigator — Sao Paulo State University - Brazil
Locations (1):
- Mauro Pedrine Santamaria and Manuela Maria Viana Miguel, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the end of the study after a direct request
Supporting Information: Study Protocol, ICF
Time Frame: After the study completion.

REFERENCES:
- [Background] Teuschl AH, Zipperle J, Huber-Gries C, Kaplan DL. Silk fibroin based carrier system for delivery of fibrinogen and thrombin as coagulant supplements. J Biomed Mater Res A. 2017 Mar;105(3):687-696. doi: 10.1002/jbm.a.35940. Epub 2016 Nov 7. PMID 27756117
- [Background] Kamalathevan P, Ooi PS, Loo YL. Silk-Based Biomaterials in Cutaneous Wound Healing: A Systematic Review. Adv Skin Wound Care. 2018 Dec;31(12):565-573. doi: 10.1097/01.ASW.0000546233.35130.a9. PMID 30475285
- [Background] Chen X, Liu Y, Zhang X. Topical insulin application improves healing by regulating the wound inflammatory response. Wound Repair Regen. 2012 May-Jun;20(3):425-34. doi: 10.1111/j.1524-475X.2012.00792.x. PMID 22564234
- [Background] Dias SB, Fonseca MV, Dos Santos NC, Mathias IF, Martinho FC, Junior MS, Jardini MA, Santamaria MP. Effect of GaAIAs low-level laser therapy on the healing of human palate mucosa after connective tissue graft harvesting: randomized clinical trial. Lasers Med Sci. 2015 Aug;30(6):1695-702. doi: 10.1007/s10103-014-1685-2. Epub 2014 Nov 6. PMID 25373688
- [Derived] Santamaria MP, Mathias-Santamaria IF, Ferreira Bonafe AC, Gonzalez OA, Kirakodu S, Monteiro MF, Casarin RCV, Shaddox LM, Miguel MMV. Microbiome and Inflammatory Biomarkers Associated With Palatal Wound Healing. J Periodontal Res. 2025 Jul;60(7):664-675. doi: 10.1111/jre.13373. Epub 2025 Jan 13. PMID 39801488